CLINICAL TRIAL: NCT00880425
Title: Do Patients With Chronic Daily Headache Have Continuous Headache or Moments of Headache Relief?
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Stephen D. Silberstein, Professor of Neurology, Thomas Jefferson University
Other Study IDs: SDS/CDH/01
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2010-10-29 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Chronic Daily Headache
MeSH Terms: conditions — Headache Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants with continuous headache
- Participants with non-continuous headache

SUMMARY:
The objective of this study is to determine if patients with chronic daily headache have continuous headache or moments of headache relief. The secondary objective of this study is to determine the period of time patients who have chronic daily headache that is not continuous are headache free.

DETAILED DESCRIPTION:
This study is a retrospective chart review of all patients over the age of 18 who are seen by the co-investigator during one initial, or routine follow up visit, with the diagnosis of chronic migraine, chronic tension type headache, new daily persistent headache, or chronic post traumatic headache(per International Headache Classification II guidelines6). Patients with the above diagnosis during their routine care are asked five standard questions about their headaches by the co-investigator, and the responses are recorded in the patient's medical record (see question sheet attached). These questions pertain to the patients' health care, and are asked of most patients at the Jefferson Headache center with chronic headache routinely during office visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Migraine, New Daily Persistent Headache, Chronic Tension type headache, or chronic post traumatic headache seen at the Jefferson Headache Center.

Exclusion Criteria:

* Subjects under age 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Headache clinic patients with diagnosis of Chronic Migraine, New Daily Persistent Headache, Chronic Tension type headache, or chronic post traumatic headache, over age 18.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Silberstein, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Jessica Ailani, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Headache Every Day (HED) Non-continuous; Headache Every Day Continuous: Subjects with Headache every day included those with a diagnosis of Chronic Migraine, New Daily Persistent Headache, Chronic Post Traumatic Headache and Chronic TensionType Headache
Period: Overall Study
Arm/Group | Headache Every Day (HED) Non-continuous | Headache Every Day Continuous
Started | 18 | 27
Completed | 18 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Chronic Daily Headache: Patients who fulfilled criteria for Chronic Migraine, New Daily Persistent Headache , Chronic Post Traumatic Headache or Chronic Tension Type Headache
Arm/Group | Chronic Daily Headache
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Daily Headache Who Have Continuous Headache
Time Frame: Records were reviewed from April 2009 through June 2009
Measure: Number; unit: participants
Arm/Group | Headache Every Day (HED) Non-continuous | Headache Every Day Continuous
Number analyzed (Participants) | 18 | 27
participants | 18 | 27

2. Secondary Outcome: Number of Patient With Daily Headache Who Have Non-continuous Headache
Time Frame: Records were reviewed from April 2009 through June 2009
Measure: Number; unit: participants
Arm/Group | Headache Every Day (HED) Non-continuous | Headache Every Day Continuous
Number analyzed (Participants) | 18 | 27
participants | 18 | 27

ADVERSE EVENTS:
Arm/Group | Headache Every Day (HED) Non-continuous | Headache Every Day Continuous
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/27
Other Adverse Events (participants affected / at risk) | 0/18 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No